CLINICAL TRIAL: NCT00830635
Title: Cancer Information Service Research Consortium: Years 2006-2011 Program Narrative and Overview
Brief Title: Multimedia Educational Program for Patients With Early-Stage Prostate Cancer or Breast Cancer
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Colorado, Denver (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None
Other Study IDs: 08-0498; AMCCRC-08-0498
Record Dates: First submitted 2009-01-27; First posted 2009-01-28 (Estimated); Last update posted 2015-06-16 (Estimated); Status verified 2015-06

CONDITIONS: Breast Cancer; Depression; Long-term Effects of Cancer Treatment; Prostate Cancer; Psychosocial Effects of Cancer and Its Treatment
Keywords: long-term effects of cancer treatment; psychosocial effects of cancer and its treatment; depression; stage IA breast cancer; stage IB breast cancer; stage II breast cancer; stage I prostate cancer; stage II prostate cancer
MeSH Terms: conditions — Breast Neoplasms; Depression; Prostatic Neoplasms | interventions — Early Intervention, Educational; Psychiatric Rehabilitation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Other: educational intervention
Other: informational intervention
Other: internet-based intervention
Other: questionnaire administration
Other: study of socioeconomic and demographic variables
Other: survey administration
Procedure: psychosocial assessment and care
Procedure: quality-of-life assessment

SUMMARY:
RATIONALE: A multimedia educational program may help patients with newly diagnosed prostate cancer and breast cancer reduce distress, make informed treatment decisions, and improve quality of life.

PURPOSE: This randomized clinical trial is studying how well a multimedia educational program works in patients with early-stage prostate cancer or breast cancer.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* Determine whether an innovative multimedia educational program will help newly diagnosed prostate (project 1) and breast (project 2) cancer patients prepare for their journey as cancer patients, promote informed treatment decision-making and reduce cancer-specific distress, and among breast cancer patients at re-entry, facilitate an informed re-entry transition to cancer survivorship and reduce cancer-specific distress (project 3).
* Determine whether having Cancer Information Service (CIS) Information Specialists make a scheduled telephone callback to callers in project 3 will augment and support use of the CIS Research Consortium (CISRC) multimedia educational programs and further enhance the study outcomes examined in this program of research.
* Determine whether the hypothesized mediational variables account for significant intervention effects in each of the three component projects.
* Examine potential moderator variables to assess potential differences in intervention efficacy by selected subgroups (e.g., age, education) within each component project.
* Conduct an in-depth tracking study of utilization patterns for a detailed description of different patterns of use, as well as elucidating those components or modules within the program that had differential utilization by participants.
* Assist the CIS and other similar cancer information systems in disseminating one or more of the CISRC interventions should they prove effective in this program of research.

Secondary

* Conduct secondary analyses across projects (i.e., perceived need for and benefit from the CISRC interventions and intervention efficacy across three high priority cancer patient populations) that will be made possible by the use of a common theoretical framework, the same or similar intervention and research design across projects, and a common set of endpoints.

OUTLINE: This is a multicenter study.

Patients are assessed by demographic questions and a baseline interview conducted by Cancer Information Service (CIS) Information Specialists.

Patients are randomized to 1 of 3 intervention groups:

* Group 1: Patients receive a mailing containing standard CIS print materials. In project 1, patients receive " Treatment Choices for Men with Early-Stage Prostate Cancer" and "What You Need to Know About Prostate Cancer". In project 2, patients receive "What You Need to Know About Breast Cancer" and "Surgery Choices for Women with Early-Stage Breast Cancer". In project 3, patients receive "Facing Forward: Life After Cancer Treatment" and "What You Need to Know About Breast Cancer".
* Group 2: Patients receive mailings appropriate to their project as in group 1. Patients also receive the multimedia program via the Internet or CD-ROM.
* Group 3: In project 3 only, patients receive mailings appropriate to their project as in group 1 and the multimedia program as in group 2. Patients also receive a CIS callback intervention at 10-14 days from trained Information Specialists from the CIS.

After completion of study therapy, patients are followed at 2 and 9 months.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Patients are diagnosed with 1 of the following:

  * Diagnosis of prostate cancer (project 1)

    * Early-stage disease
    * Previously untreated disease or treatment status unknown
  * Diagnosis of breast cancer (projects 2-3)

    * Early-stage disease
    * No ductal carcinoma in situ or lobular carcinoma in situ
    * Inflammatory breast cancer allowed (project 2)
    * Previously untreated disease, receiving concurrent treatment, previously treated disease, or treatment status unknown

      * No more than 30 days since completion of treatment OR no more than 6 months post-treatment (project 3)

PATIENT CHARACTERISTICS:

* Has access to a computer
* Willing to provide mailing address and telephone number
* Must be active information-seekers who have already called the CIS
* Understands English

PRIOR CONCURRENT THERAPY:

* See Disease Characteristics

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 1800 (Actual)
Dates: Start 2008-09; Primary Completion 2013-04 (Actual); Study Completion 2013-12 (Actual)

PRIMARY OUTCOMES:
Cancer-specific distress
Emotional quality of life
Physical functioning
Interpersonal functioning
Benefit-finding
Decisional conflict (projects 1 and 2)
Regret (projects 1 and 2)
Fear of recurrence (project 3)
Practical concerns (project 3)

CONTACTS AND LOCATIONS:
Overall Officials: Alfred Marcus, PhD, Principal Investigator — AMC Cancer Research Center
Locations (3):
- United States (3):
  - University of Miami Sylvester Comprehensive Cancer Center - Miami, Miami, Florida
  - Memorial Sloan-Kettering Cancer Center, New York, New York
  - Fred Hutchinson Cancer Research Center, Seattle, Washington